CLINICAL TRIAL: NCT02534909
Title: An Open-label Proof of Concept Study to Assess the Efficacy, Safety and Pharmacokinetics of LFG316, an Anti-C5 Monoclonal Antibody in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Proof of Concept Study to Assess the Efficacy, Safety and Pharmacokinetics of LFG316 in Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLFG316X2201; 2014-005338-74 (EudraCT Number)
Record Dates: First submitted 2015-08-07; First posted 2015-08-28 (Estimated); Results first posted 2024-11-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria (PNH); LFG316; LNP023
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Intervention Model Description: All patients were on active treatment.
  In treatment periods 1 to 3, patients received the following:
  • LFG316 20 mg/kg as i.v. infusion every 2 weeks
  Patients participating in treatment period 4 received the following:
  * LFG316 20 mg/kg as i.v. infusion every 2 weeks for 4 weeks (total 2 infusions)
  * LNP023 200 mg b.i.d. for approximately 20 weeks. Four capsules (each 50 mg) were administered each time study medication was taken.
  Down-titration was permitted only in case of LNP023 treatment discontinuation:
  * LNP023 30 mg taken in the evening (once daily) for 7 days (3 capsules of 10 mg each time study medication was taken).
  * Followed by LNP023 10 mg taken in the evening (once daily) for 7 days (1 capsule of 10 mg each time study medication was taken).
  * LFG316 was administered via i.v. infusion by the investigator or designated study staff over approximately 2 hours in Period 1 and between 40 minutes and 2 hours from Period 2 onwards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LFG316 then LNP023 (Experimental): During treatment periods 1 to 3, the regimen included LFG316 at a dosage of 20 mg/kg administered as an intravenous (i.v.) infusion biweekly.
  In treatment period 4, the patients were given:
  * LFG316 at a dosage of 20 mg/kg as an i.v. infusion every two weeks for four weeks, amounting to two infusions in total.
  * LNP023 at a dose of 200 mg administered orally twice daily (b.i.d.) for approximately 20 weeks, with four 50 mg capsules taken at each administration.
  Interventions: Biological: LFG316; Drug: LNP023

INTERVENTIONS:
Biological: LFG316 — LFG316 20 mg/kg was administered to all patients enrolled in the study:
  * Treatment Periods 1 to 3: LFG316 20 mg/kg as i.v. infusion every 2 weeks
  * Treatment Period 4: LFG316 20 mg/kg as i.v. infusion every 2 weeks for 4 weeks (total 2 infusions).
Drug: LNP023 — Treatment Period 4: LNP023 200 mg b.i.d. for approximately 20 weeks. Four capsules (each 50 mg) were administered each time study medication was taken.

SUMMARY:
The purpose of this study was to determine whether LFG316 can induce a hematological response, as measured by reduction in hemolytic activity, in patients with paroxysmal nocturnal hemoglobinuria (PNH).

DETAILED DESCRIPTION:
The study consisted of a 60-day screening period to assess eligibility and conduct vaccinations if required (for all patients not previously vaccinated at least 2 weeks prior to first dosing or if prior vaccination cannot be confirmed) and 4 treatment periods as follows. During the treatment period 1 (Days 1 to 29), all patients received infusions of LFG316 every 14 days. Following assessment of efficacy (hemolytic activity by serum LDH) at the end of treatment period 1, patients entered the optional 48-week treatment period 2 and continued LFG316 infusions every 14 days. At the end of treatment period 2, LFG316-responsive patients (assessed based on the investigator's judgment) were allowed to enter an additional extension period of up to 260 weeks (treatment period 3) in which they continued to receive LFG316 every 14 days. Period 4, which allowed patients to switch to LNP023, lasted approximately 21 weeks. During the first 4 weeks, patients continued to receive LFG316 in addition to oral administration of LNP023. After 4 weeks, patients discontinued LFG316 and continued with LNP023 monotherapy for approximately 16 weeks (+/- 28 days). Patients who participated in period 4 could join the long-term extension study CLNP023C12001B (NCT04747613) as soon as their eligibility was confirmed and study CLNP023C12001B was open to receive patients. There was no LNP023 treatment gap between the studies.

As per strategic decision, further development of LFG316 was terminated in favor of LNP023, Novartis offered patients enrolled in study CLFG316X2201 a conversion from LFG316 to LNP023, aiming to provide uninterrupted treatment for these PNH patients. The CLFG316X2201 trial was not a terminated study.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent obtained before any assessment were performed.
2. Male and female patients >= 18 years old with a diagnosis of PNH prior to screening. Based on local requirements (applicable in Czech Republic) only patients between the age of 18 to 65 (inclusive) with a diagnosis of PNH prior to screening were eligible for inclusion in this study.
3. A documented PNH clone size of >= 10% by RBCs and/or granulocytes, measured by GPI deficiency on flow cytometry.
4. Serum LDH levels at least 1.5-fold above the ULN at screening.
5. Patients receiving treatment with corticosteroids and/or other immunosuppressive regimens could continue treatment throughout the study, if indicated for treatment of autoimmune disease (e.g., aplastic anemia). It was strongly recommended, at the investigator's discretion, that patients receive appropriate prophylactic antibiotics (e.g., ciprofloxacin, penicillin, erythromycin) while on treatment with any type of concomitant immunosuppressive agent other than LFG316 (including corticosteroids).
6. Negative pregnancy test for women of child-bearing potential at screening.
7. Previous vaccination against Neisseria meningitidis types A, C, Y and W-135 at least 2 weeks prior to first dosing, and vaccination against meningitidis type B if available and acceptable by local regulations, at least 2 weeks prior to first dosing.
8. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

   Patients included in this study after protocol amendment 6 were also to fulfill the following:
9. To be carriers of the C5 gene minor variants as defined by nucleic acid changes that lead to amino acid exchanges in position p.Arg885.

   Additional inclusion criteria for period 4
10. Patients who participated in period 3 of the current study who wanted to join the long-term extension study with LNP023 (CLNP023C12001B).
11. Previous vaccination for the prevention of Streptococcus pneumoniae and Haemophilus influenzae at least 2 weeks prior to first dosing with LNP023 if locally available. If LNP023 treatment had to start earlier than 2 weeks post vaccination, prophylactic antibiotic treatment was required.

Exclusion criteria:

1. Known or suspected hereditary complement deficiency.
2. History of hematopoietic stem cell transplantation.
3. Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedure within 30 days or 5-times the half-life prior to screening. Note: clinical trials solely involving over-the-counter vitamins, off label use of drugs within published standard of care guidelines, supplements, or diet did not exclude an otherwise eligible patient.
4. Female patients who were pregnant, breastfeeding, or intended to conceive during the course of the study.
5. History of recurrent meningitis, history of meningococcal meningitis despite vaccination.
6. Presence or suspicion (based on judgment of the investigator) of severe active bacterial infection within 2 weeks prior to first dose of LFG316, or severe recurrent bacterial infections.
7. A positive HIV test result.
8. Under active therapy with other agents interfering with the complement system (e.g., eculizumab) Wash-out time was at least 5 half-lives, approximately 8 weeks for eculizumab.
9. Severe concurrent co-morbidities, e.g., patients with severe kidney disease (dialysis), advanced cardiac disease (NYHA class IV), severe pulmonary arterial hypertension (WHO class IV), unstable thrombotic event not amenable to active treatment as judged by the investigator.
10. Either one of the following laboratory abnormalities at screening:

    * Neutrophils < 0.5 × 10^9/L
    * Platelets < 30 × 10^9/L
11. Co-morbidities that were likely caused by underlying autoimmune diseases other than PNH, e.g., kidney disease in the context of lupus nephritis, ANCA-associated vasculitis.
12. Any medical condition deemed likely to interfere with the patient's participation in the study, or likely to cause serious adverse events during the study.
13. History of hypersensitivity to a drug of the same class (human IgG1 monoclonal antibody) or any other excipient of the formulation.
14. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using highly effective methods of contraception during dosing and for 50 days after the last dose of LFG316.
15. Prohibited medication as specified in the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Brno-Bohunice, Czech Republic, Czechia
- Japan (5):
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Niigata
- Novartis Investigative Site, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 participants were enrolled at 7 sites in 3 countries.
Pre-assignment Details: The study had a 60-day screening period to assess eligibility.
Groups:
- LFG316 Then LNP023: Treatment periods 1 to 3: LFG316 20 mg/kg intravenous (i.v.) infusion every 2 weeks.
  Treatment period 4: LFG316 20 mg/kg intravenous (i.v.) infusion every 2 weeks (Week 1 to 4) + LNP023 200 mg twice per day (b.i.d.) for approximately 20 weeks (Weeks 1 to 20)
Period: Treatment Period 1 to 3 (up to Week 312)
Arm/Group | LFG316 Then LNP023
Started (All enrolled patients were included in the Safety and Pharmacokinetic (PK) analysis sets) | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Treatment Period 4 (20 Weeks)
Arm/Group | LFG316 Then LNP023
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LFG316 Then LNP023
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3
  Asian | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reduction in Serum Lactate Dehydrogenase (LDH) Levels Within the First 4 Weeks of LFG316 Treatment as Measured by Response Rate
Description: The primary efficacy variable for assessing the effect of LFG316 over the first 4 weeks of treatment was response rate where a patient was considered a responder if the percentage reduction from baseline in serum lactate dehydrogenase (LDH) was at least 60% at any time up to and including week 4 for that patient.
Time Frame: Overall (Up to Week 4), Period 1 Day 8, Period 1 Day 15, Period 1 Day 22, Period 1 Day 29
Population: The Pharmacodynamic (PD) analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Count of Participants; unit: Participants
Arm/Group | LFG316 Then LNP023
Number analyzed (Participants) | 10
Participants
  Overall (Up to Week 4): Responder | 10
  Overall (Up to Week 4): Non Responder | 0
  Period 1 Day 8: Responder | 6
  Period 1 Day 8: Non Responder | 4
  Period 1 Day 15: Responder | 9
  Period 1 Day 15: Non Responder | 1
  Period 1 Day 22: Responder | 9
  Period 1 Day 22: Non Responder | 1
  Period 1 Day 29: Responder | 9
  Period 1 Day 29: Non Responder | 1
Statistical Analysis 1: Comparison: LFG316 Then LNP023; Up to Week 4; Test type: Other — Bayesian analysis of response rate in serum LDH (period 1 completers only); Median response rate = 99.0, 95% CI 2-sided [81.9 to 100.0] — 95% Credibility Interval for Response Rate

2. Primary Outcome: Percentage Change From Baseline in Serum Lactate Dehydrogenase (LDH) Levels Over the Entire Treatment Period
Description: Lactate dehydrogenase (LDH) levels were measured in serum samples and the percentage change from baseline was calculated. For serum LDH, baseline was the average of all pre-dose measurements.
Time Frame: Baseline, Period 1 Day 29 (end of Treatment Period 1), Period 2 Day 365 (end of Treatment Period 2), Period 3 Day 1429 (end of Treatment Period 3), Period 4 Day 141 (end of Treatment Period 4)
Population: Pharmacodynamic (PD) analysis set - Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: % change from baseline in serum LDH
Arm/Group | LFG316 Then LNP023
Number analyzed (Participants) | 10
% change from baseline in serum LDH
  Period 1 Day 29 | -78.35 (11.190)
  Period 2 Day 365 | -78.56 (11.550)
  Period 3 Day 1429 | -81.65 (8.138)
  Period 4 Day 141: number analyzed (Participants) | 9
  Period 4 Day 141 | -78.69 (9.288)
Statistical Analysis 1: Comparison: LFG316 Then LNP023; Period 1 Day 29 serum LDH levels; Test type: Other; p < 0.001, Mixed Models Analysis; Geometric LS mean Ratio to Baseline = 0.19, 95% CI 2-sided [0.15 to 0.23] — The longitudinal mixed effects model included timepoint, log baseline as a covariate and the log baseline by timepoint interaction. C5 variant status was included as a categorical covariate
Statistical Analysis 2: Comparison: LFG316 Then LNP023; Period 2 Day 365 serum LDH levels; Test type: Other; p < 0.001, Mixed Models Analysis; Geometric LS mean Ratio to Baseline = 0.19, 95% CI 2-sided [0.15 to 0.23] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: LFG316 Then LNP023; Period 3 Day 1429 serum LDH levels; Test type: Other; p < 0.001, Mixed Models Analysis; Geometric LS mean Ratio to Baseline = 0.17, 95% CI 2-sided [0.14 to 0.20] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: LFG316 Then LNP023; Period 4 Day 141 serum LDH levels; Test type: Other; p < 0.001, Mixed Models Analysis; Geometric LS mean Ratio to Baseline = 0.19, 95% CI 2-sided [0.15 to 0.24] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to the Last Measurable Serum Concentration Sampling Time (0-tlast) for LFG316
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization of LFG316. Pharmacokinetic parameters were determined using non-compartmental methods based on LFG316 concentrations in serum. AUC (0-tlast) was summarized using descriptive statistics.
Time Frame: Pre-infusion and 2 hours after the end of infusion on Period 1 Day 1.
Population: Pharmacokinetic (PK) analysis set included all patients with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: hour*microgram/milliliter (h*µg/mL)
Arm/Group | LFG316 Then LNP023
Number analyzed (Participants) | 10
hour*microgram/milliliter (h*µg/mL) | 73700 (12600)

4. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for LFG316
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization of LFG316. Pharmacokinetic parameters were determined using non-compartmental methods based on LFG316 concentrations in serum. Cmax was summarized using descriptive statistics.
Time Frame: Pre-infusion and 2 hours after the end of infusion on Period 1 Day 1.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (μg/mL)
Arm/Group | LFG316 Then LNP023
Number analyzed (Participants) | 10
nanograms per milliliter (μg/mL) | 407 (69.2)

5. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) for LFG316
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization of LFG316. Pharmacokinetic parameters were determined using non-compartmental methods based on LFG316 concentrations in serum. Tmax was summarized using descriptive statistics. Actual sampling times were used for the calculation of PK parameters.
Time Frame: Pre-infusion and 2 hours after the end of infusion on Period 1 Day 1.
Population: PK analysis set
Measure: Median (Full Range); unit: hour (h)
Arm/Group | LFG316 Then LNP023
Number analyzed (Participants) | 10
hour (h) | 2.56 [2.05 to 3.10]

6. Secondary Outcome: LFG316 Serum Concentration
Description: The concentration of total LFG316 in serum was determined using Liquid chromatography/mass spectroscopy (LC/MS assay) and summarized using descriptive statistics.
Time Frame: Period 1 Day 1 (predose (trough), post-dose), Period 2 Day 337 (predose), Period 3 Day 1289 (predose)
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (μg/mL)
Arm/Group | LFG316 Then LNP023
Number analyzed (Participants) | 10
nanograms per milliliter (μg/mL)
  Period 1 Day 1 (predose (trough)) | 182 (31.4)
  Period 1 Day 1 (postdose) | 538 (80.0)
  Period 2 Day 337 (predose) | 248 (55.9)
  Period 3 Day 1289 (predose) | 313 (89.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of LFG316 (Day 1) up to 4 weeks after last dose (Day 2213) in participants transitioning to Period 4 and up to 8 weeks after last dose (Day 2241) in participants ending participation after Period 3. In Period 4, adverse events were collected from first dose of study treatment (Day 1) up to approximately 30 days after last dose of LNP023 (Day 171).
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Groups:
- Treatment Periods 1 to 3: LFG316: Treatment Periods 1 to 3: LFG316 20 mg/kg intravenous (i.v.) infusion every 2 weeks.
- Treatment Period 4: LFG316 + LNP023: Treatment Period 4: LFG316 20 mg/kg intravenous (i.v.) infusion every 2 weeks (Week 1 to 4) + LNP023 200 mg twice per day (b.i.d.) for approximately 20 weeks (Weeks 1 to 20)
Arm/Group | Treatment Periods 1 to 3: LFG316 | Treatment Period 4: LFG316 + LNP023
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/9
Other Adverse Events (participants affected / at risk) | 10/10 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Periods 1 to 3: LFG316 (N=10) | Treatment Period 4: LFG316 + LNP023 (N=9)
Bacteraemia (Infections and infestations) | 1 | 0
Enterocolitis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Periods 1 to 3: LFG316 (N=10) | Treatment Period 4: LFG316 + LNP023 (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Brugada syndrome (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Immunisation reaction (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Helicobacter infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 0
Lyme disease (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 0
Paronychia (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0
International normalised ratio decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 5 | 1
Migraine (Nervous system disorders) | 2 | 0
Migraine with aura (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT02534909/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT02534909/SAP_001.pdf